CLINICAL TRIAL: NCT02808845
Title: Pre-existing Microalbuminuria Predicting Contrast-induced Acute Kidney Injury (CIAKI) Following Coronary Angiography (CAG)
Brief Title: Microalbuminuria Predicting CIAKI After CAG
Acronym: MPCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CIAKI-1
Record Dates: First submitted 2016-06-13; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Contrast-induced Acute Kidney Injury; Microalbuminuria
Keywords: coronary angiography; contrast-induced acute kidney injury; microalbuminuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- microalbuminuria with eGFR≥60ml/min: microalbuminuria group with estimated glomerular filtration rate (eGFR) ≥60ml/min.
  Interventions: Other: microalbuminuria
- normal-albuminuria group with eGFR≥60ml/min: normal-albuminuria group with estimated glomerular filtration rate (eGFR) ≥60ml/min.
- microalbuminuria group with eGFR<60ml/min: microalbuminuria group with estimated glomerular filtration rate (eGFR) <60ml/min.
  Interventions: Other: microalbuminuria
- normal-albuminuria group with eGFR<60ml/min: normal-albuminuria group with estimated glomerular filtration rate (eGFR) <60ml/min.

INTERVENTIONS:
Other: microalbuminuria
  Groups: microalbuminuria group with eGFR<60ml/min; microalbuminuria with eGFR≥60ml/min

SUMMARY:
The purpose of this study is to investigate the association between pre-existing microalbuminuria and contrast-induced acute kidney injury (CIAKI) following coronary angiography (CAG).

ELIGIBILITY:
Inclusion Criteria:

* Patients with eGFR≥30ml/min and without macroalbuminuria undergoing CAG.

Exclusion Criteria:

* Pregnancy
* Lactation
* Allergic history of contrast media
* Having been received contrast media within 7 days
* Use of nephrotoxic medications within 7 days
* eGFR <30 ml/min, macroalbuminuria (ACR >300 mg/g)
* Renal transplantation, emergent coronary angiography
* Cardiogenic shock, pulmonary edema
* Use of intra-aortic balloon pump (IABP) or mechanical ventilation
* Multiple myeloma and other malignant tumor
* Life expectancy less than 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with eGFR ≥ 30 ml/min and without macroalbuminuria (defined as urine albumin to creatinine ratio (ACR) >300 mg/g) on admission are prepared to accept scheduled invasive coronary angiography during hospitalization.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
changes of serum creatinine (SCr, umol/L) | 24-48 hours after CAG
  the difference of SCr before and after CAG.
number of participants with increase in SCr of at least 44.2 umol/L higher than before | 24-48 hours after CAG
  number of participants with the difference of SCr before and after CAG over 44.2 umol/L.
number of participants with increase of SCr over 25% higher than before | 24-48 hours after CAG
  number of participants with an increase of SCr over 25% higher than before.

SECONDARY OUTCOMES:
changes of urine albumin to creatinine ratio (ACR, mg/g) | 24-48 hours after CAG
  the difference of ACR before and after CAG

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Yang, Doctor, Study Chair — First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Pucelikova T, Dangas G, Mehran R. Contrast-induced nephropathy. Catheter Cardiovasc Interv. 2008 Jan 1;71(1):62-72. doi: 10.1002/ccd.21207. PMID 17975790
- [Background] Jo SH, Youn TJ, Koo BK, Park JS, Kang HJ, Cho YS, Chung WY, Joo GW, Chae IH, Choi DJ, Oh BH, Lee MM, Park YB, Kim HS. Renal toxicity evaluation and comparison between visipaque (iodixanol) and hexabrix (ioxaglate) in patients with renal insufficiency undergoing coronary angiography: the RECOVER study: a randomized controlled trial. J Am Coll Cardiol. 2006 Sep 5;48(5):924-30. doi: 10.1016/j.jacc.2006.06.047. Epub 2006 Aug 17. PMID 16949481
- [Background] Marenzi G, Assanelli E, Campodonico J, Lauri G, Marana I, De Metrio M, Moltrasio M, Grazi M, Rubino M, Veglia F, Fabbiocchi F, Bartorelli AL. Contrast volume during primary percutaneous coronary intervention and subsequent contrast-induced nephropathy and mortality. Ann Intern Med. 2009 Feb 3;150(3):170-7. doi: 10.7326/0003-4819-150-3-200902030-00006. PMID 19189906
- [Background] Rihal CS, Textor SC, Grill DE, Berger PB, Ting HH, Best PJ, Singh M, Bell MR, Barsness GW, Mathew V, Garratt KN, Holmes DR Jr. Incidence and prognostic importance of acute renal failure after percutaneous coronary intervention. Circulation. 2002 May 14;105(19):2259-64. doi: 10.1161/01.cir.0000016043.87291.33. PMID 12010907
- [Background] Cronin RE. Contrast-induced nephropathy: pathogenesis and prevention. Pediatr Nephrol. 2010 Feb;25(2):191-204. doi: 10.1007/s00467-009-1204-z. Epub 2009 May 15. PMID 19444480
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Lambers Heerspink HJ, Brinkman JW, Bakker SJ, Gansevoort RT, de Zeeuw D. Update on microalbuminuria as a biomarker in renal and cardiovascular disease. Curr Opin Nephrol Hypertens. 2006 Nov;15(6):631-6. doi: 10.1097/01.mnh.0000247496.54882.3f. PMID 17053479
- [Background] Stehouwer CD, Smulders YM. Microalbuminuria and risk for cardiovascular disease: Analysis of potential mechanisms. J Am Soc Nephrol. 2006 Aug;17(8):2106-11. doi: 10.1681/ASN.2005121288. Epub 2006 Jul 6. PMID 16825333
- [Background] Baber U, Mann D, Shimbo D, Woodward M, Olin JW, Muntner P. Combined role of reduced estimated glomerular filtration rate and microalbuminuria on the prevalence of peripheral arterial disease. Am J Cardiol. 2009 Nov 15;104(10):1446-51. doi: 10.1016/j.amjcard.2009.06.068. PMID 19892066
- [Background] Bakris GL, Ruilope L, Locatelli F, Ptaszynska A, Pieske B, de Champlain J, Weber MA, Raz I. Treatment of microalbuminuria in hypertensive subjects with elevated cardiovascular risk: results of the IMPROVE trial. Kidney Int. 2007 Oct;72(7):879-85. doi: 10.1038/sj.ki.5002455. Epub 2007 Aug 1. PMID 17667984
- [Background] Sany D, Refaat H, Elshahawy Y, Mohab A, Ezzat H. Frequency and risk factors of contrast-induced nephropathy after cardiac catheterization in type II diabetic patients: a study among Egyptian patients. Ren Fail. 2014 Mar;36(2):191-7. doi: 10.3109/0886022X.2013.843400. Epub 2013 Oct 21. PMID 24138570
- [Result] Meng H, Wu P, Zhao Y, Xu Z, Wang ZM, Li C, Wang L, Yang Z. Microalbuminuria in patients with preserved renal function as a risk factor for contrast-Induced acute kidney injury following invasive coronary angiography. Eur J Radiol. 2016 Jun;85(6):1063-7. doi: 10.1016/j.ejrad.2016.03.010. Epub 2016 Mar 16. PMID 27161053
- See also: Click here for more information about this study: Microalbuminuria Predicting CIAKI After CAG — http://link.springer.com/article/10.1007%2Fs00467-009-1204-z
- See also: Click here for more information about this study: Microalbuminuria Predicting CIAKI After CAG — http://linkinghub.elsevier.com/retrieve/pii/S0272638602093563
- See also: Click here for more information about this study: Microalbuminuria Predicting CIAKI After CAG — http://journals.lww.com/co-nephrolhypertens/pages/articleviewer.aspx?year=2006&issue=11000&article=00014&type=abstract
- See also: Click here for more information about this study: Microalbuminuria Predicting CIAKI After CAG — http://jasn.asnjournals.org/content/17/8/2106.long